CLINICAL TRIAL: NCT02479698
Title: Phase II Study Assessing the Effect of BK Specific CTL Lines Generated by Ex Vivo Expansion in Patients With BK Virus Infection and JC Virus Infection
Brief Title: Cytotoxic T Lymphocytes in Treating Patients With Malignancies With BK and/or JC Virus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0279; NCI-2015-01264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0279 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Acquired Immunodeficiency Syndrome; BK Virus Infection; Human Immunodeficiency Virus; JC Virus Infection; Malignant Neoplasm; Merkel Cell Carcinoma; Merkel Cell Polyomavirus Infection; Viral Encephalitis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neoplasms; Carcinoma, Merkel Cell; Encephalitis, Viral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (BK-specific cytotoxic T lymphocytes) (Experimental): Patients receive allogeneic BK-specific cytotoxic T-lymphocytes IV over 30 minutes. Patients achieving partial response, stable disease, or progressive disease are eligible for 19 additional infusions of CTL occurring at least 2 weeks after the previous CTL infusion if they meet the eligibility criteria for subsequent therapy.
  Interventions: Biological: Allogeneic BK-specific Cytotoxic T-lymphocytes; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Allogeneic BK-specific Cytotoxic T-lymphocytes — Given IV
  Other Names: Allogeneic BK-CTLs; Allogeneic BK-specific CTLs
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well donor cytotoxic T lymphocytes work in treating patients with malignancies with BK and/or JC virus. Cytotoxic T lymphocytes are made from donated blood cells that are grown in the laboratory and are designed to kill viruses that can cause infections in transplant patients and may be an effective treatment in patients with malignancies with BK and/or JC virus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy, feasibility and safety of administering most closely human leukocyte antigen (HLA)-matched BK specific cytotoxic T lymphocyte (CTL) lines (BK-CTLs) generated by ex vivo expansion to mediate antiviral activity in patients with any type of malignancies, and/or human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDs), and/or history of solid organ transplant with BK and JC infections.

SECONDARY OBJECTIVE:

I. To assess the persistence of the administered BK-CTLs generated by ex vivo expansion in patients with any type of malignancies, and/or HIV/AIDs, and/or history of solid organ transplant with BK and JC infections.

OUTLINE:

Patients receive allogeneic BK-specific cytotoxic T-lymphocytes intravenously (IV) over 30 minutes. Patients achieving partial response, stable disease, or progressive disease are eligible for 7 additional infusions of CTL occurring at least 2 weeks after the previous CTL infusion if they meet the eligibility criteria for subsequent therapy.

After completion of study treatment, patients are followed up periodically for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 2 years. English and non-English speaking patients are eligible.
* Immunocompromised patients; and/or Non-immunocompromised patients with PML/JC virus Encephalitis; and/or patients with any type of malignancies; and/or HIV/AIDs; and/or history of solid organ transplant; and/or Merkel polyoma-virus related Merkel cell tumor(s) with measurable disease on imaging per RECIST criteria.
* Patients with microscopic hematuria OR biopsy proven BK nephritis and urine or blood PCR positive for BK virus and/or JC viral encephalitis and/or JC end-organ disease and/or polyomavirus.
* Clinical status at enrollment to allow tapering of steroids to less than 0.5 mg/kg/day of prednisone.
* Patients who are currently receiving treatment with cidofovir, leflunomide, or other antiviral therapy with no response, will be eligible for CTL infusion.
* Written informed consent and/or signed assent from patient, parent or guardian. Patients with cognitive impairments are eligible.
* Negative pregnancy test in female patients of childbearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization. Women of child bearing potential must be willing to use an effective contraceptive measure while on study.
* Patients enrolled on this study may be enrolled on other IND studies at the discretion of the PI.
* Patients may be re-enrolled in the protocol should the infection re-occur, provided they meet all the other eligibility criteria at the moment of re-enrollment.

Exclusion Criteria:

* Patients receiving prednisone > 0.5 mg/kg/day at time of enrollment, or have received ATG within 14 days or have received donor lymphocyte infusion (DLI) or Campath within 28 days of enrollment.
* Patients with other uncontrolled infections (except HIV/AIDS). For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection
* Patients with active acute (GVHD) grades II-IV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07-23 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Response, defined as response (R) = (best response [R1] or second best response [R2]) | Up to 56 days
  The method of Thall et al will be used to monitor the probabilities of response.
Incidence of acute graft-versus-host disease (GVHD) | Within 28 days of the last dose of cytotoxic T lymphocytes (CTLs)
  The method of Thall et al will be used to monitor the probabilities of grade 3 or 4 GVHD.
Incidence of adverse events | Up to day 100
  Will be continuously monitored.

SECONDARY OUTCOMES:
Overall survival | Up to 12 months
  Each outcome will be evaluated by tabulation and by fitting a Bayesian statistical regression model for binary outcomes as a function of covar. Unadjusted event time distributions will be estimated using the Kaplan-Meier method.
Glomerular filtration rate | Up to 12 months
  Each outcome will be evaluated by tabulation and by fitting a Bayesian statistical regression model for binary outcomes as a function of covar. Unadjusted event time distributions will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Olson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Olson A, Lin R, Marin D, Rafei H, Bdaiwi MH, Thall PF, Basar R, Abudayyeh A, Banerjee P, Aung FM, Kaur I, Abueg G, Rao S, Chemaly R, Mulanovich V, Al-Atrash G, Alousi AM, Andersson BS, Anderlini P, Bashir Q, Castro KM, Daher M, Galvan IM, Hosing C, Im JS, Jones RB, Kebriaei P, Khouri I, Mehta R, Molldrem J, Nieto Y, Oran B, Popat U, Qazilbash M, Rondon G, Saini N, Spencer B, Srour S, Washington D, Barnett M, Champlin RE, Shpall EJ, Rezvani K. Third-Party BK Virus-Specific Cytotoxic T Lymphocyte Therapy for Hemorrhagic Cystitis Following Allotransplantation. J Clin Oncol. 2021 Aug 20;39(24):2710-2719. doi: 10.1200/JCO.20.02608. Epub 2021 Apr 30. PMID 33929874
- [Derived] Muftuoglu M, Olson A, Marin D, Ahmed S, Mulanovich V, Tummala S, Chi TL, Ferrajoli A, Kaur I, Li L, Champlin R, Shpall EJ, Rezvani K. Allogeneic BK Virus-Specific T Cells for Progressive Multifocal Leukoencephalopathy. N Engl J Med. 2018 Oct 11;379(15):1443-1451. doi: 10.1056/NEJMoa1801540. PMID 30304652
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org